CLINICAL TRIAL: NCT05476926
Title: Real-World, Long-Term Data Collection to Gain Clinical Insights Into Roche Ophthalmology Products (VOYAGER STUDY)
Brief Title: A Real-World Study to Gain Clinical Insights Into Roche Ophthalmology Products
Acronym: VOYAGER
Status: Active, not recruiting | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: MR41927
Record Dates: First submitted 2022-07-25; First posted 2022-07-27 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Neovascular Age-related Macular Degeneration; Diabetic Macular Edema; Retinal Vein Occlusion; Branch Retinal Vein Occlusion; Central Retinal Vein Occlusion; Hemi-retinal Vein Occlusion
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — faricimab; Ranibizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (5):
- Cohort 1: Faricimab for nAMD
  Interventions: Drug: Faricimab
- Cohort 2: Faricimab for DME
  Interventions: Drug: Faricimab
- Cohort 3: Port Delivery System with Ranibizumab for nAMD
  Interventions: Combination Product: Port Delivery System with Ranibizumab
- Cohort 4: Faricimab for BRVO
  Interventions: Drug: Faricimab
- Cohort 5: Faricimab for CRVO/HRVO
  Interventions: Drug: Faricimab

INTERVENTIONS:
Drug: Faricimab — Faricimab will be administered as per local clinical practice and local labeling.
  Other Names: VABYSMO™; RO6867461; RG7716
  Groups: Cohort 1: Faricimab for nAMD; Cohort 2: Faricimab for DME; Cohort 4: Faricimab for BRVO; Cohort 5: Faricimab for CRVO/HRVO
Combination Product: Port Delivery System with Ranibizumab — The port delivery system with ranibizumab will be administered as per local clinical practice and local labeling.
  Other Names: SUSVIMO™; RG6321
  Groups: Cohort 3: Port Delivery System with Ranibizumab for nAMD

SUMMARY:
The VOYAGER study is a primary data collection, non-interventional, prospective, multinational, multicenter study. It is designed to collect real-world, long-term data to explore long-term effectiveness, safety, clinical insights, treatment patterns, and factors driving the treatment decisions among patients being treated with specified Roche ophthalmology products in approved retinal indications (Faricimab for neovascular age-related macular degeneration [nAMD], diabetic macular edema [DME], and retinal vein occlusion; Port Delivery System with Ranibizumab for nAMD) in routine clinical practice. This study will not provide or make recommendations on use of any products including Roche products; treatment decisions will be determined by the treating physician and must be made independently to the decision to participate in this study. Participation in this study will not change or influence a patient's standard of care in any way.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided informed consent, as required per local regulations 2.a) Adult patient, as defined by local regulations and local product label, who is newly initiating treatment (or initiated treatment in the previous visit) with a specified approved Roche ophthalmology product in retinal indication of interest for this study in at least one eye, according to the investigator's discretion in routine clinical practice; OR 2.b) Adult patient, as defined by local regulations and local product label, who is continuing treatment with any specified approved Roche ophthalmology product in retinal indication of interest for this study in at least one eye after initiating that treatment in a Roche interventional trial.

Exclusion Criteria:

1. Concomitant participation of the patient in an investigational ophthalmology clinical trial that includes receipt of any investigational drug or procedure within the last 28 days prior to enrollment (this restriction does not apply to patients who are rolling over from Roche interventional studies and continuing treatment with any specified approved Roche ophthalmology product in retinal indication of interest for this study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients being treated with specified Roche ophthalmology products approved in retinal indications in real-world, routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Visual Acuity from Baseline at 1 Year, per Approved Retinal Indication and Product | Baseline and 1 year
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.

SECONDARY OUTCOMES:
Change in Visual Acuity from Baseline Over Time, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.
Percentage of Eyes on Each Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other) Over Time, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
Number of Treatments Over Time, per Approved Retinal Indication and Product | At 3, 6, and 12 months, and annually thereafter (up to 5 years)
Cumulative Time Spent on Each Treatment per Eye, Overall and per Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other), per Approved Retinal Indication and Product | From Baseline until end of study (up to 5 years)
Percentage of Eyes with Treatment Switch by Reason for Switch Over Time, per Approved Retinal Indication and Product | At 3, 6, and 12 months, and annually thereafter (up to 5 years)
Percentage of Eyes with Treatment Regimen Switch (Fixed, Treat-and-Extend, As Needed, or Other) by Reason for Switch Over Time, per Approved Retinal Indication and Product | At 3, 6, and 12 months, and annually thereafter (up to 5 years)
Total Number of Visits per Year, per Approved Retinal Indication and Product | Annually (up to 5 years)
Number of Visits With or Without Treatment per Year, per Approved Retinal Indication and Product | Annually (up to 5 years)
Time Interval Between Treatments per Year, per Approved Retinal Indication and Product | Annually (up to 5 years)
Number of Eyes Treated with Ocular Concomitant and Subsequent Medications by Type and Frequency During the Study, per Approved Retinal Indication and Product | From Baseline until end of study (up to 5 years)
Change in Visual Acuity from Baseline Over Time, According to Treatment Regimen (Fixed, Treat-and-Extend, As Needed, or Other), per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.
Change in Visual Acuity from Baseline Over Time, According to Number of Treatments, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.
Change in Visual Acuity from Baseline Over Time, According to Total Number of Visits, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.
Change in Visual Acuity from Baseline Over Time, According to Treatment Schedule, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
  Visual acuity will be collected as measured per local practice and then will be converted to the approximate ETDRS letter score.
Change in Central Subfield Thickness (CST) from Baseline Over Time, per Approved Retinal Indication and Product | Baseline, 3, 6, and 12 months, and annually thereafter (up to 5 years)
Number of Participants with at Least One Ocular Adverse Event, by Severity and Seriousness, per Approved Retinal Indication and Product | From Baseline until end of study (up to 5 years)
  Severity and seriousness will be independently assessed for each adverse event (AE). The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (e.g., rated as mild, moderate, or severe); the event itself may be of relatively minor medical significance.
Number of Participants with at Least One Non-Ocular Adverse Event, by Severity and Seriousness, per Approved Retinal Indication and Product | From Baseline until end of study (up to 5 years)
  Severity and seriousness will be independently assessed for each adverse event (AE). The terms "severe" and "serious" are not synonymous. Severity refers to the intensity of an AE (e.g., rated as mild, moderate, or severe); the event itself may be of relatively minor medical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (296):
- United States (18):
  - Retinal Research Institute, LLC, Phoenix, Arizona
  - California Eye Specialists Medical group Inc., Pasadena, California
  - Retinal Consultants Medical Group, Sacramento, California
  - Advanced Research, Coral Springs, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - University Retina and Macula Associates, PC, Lemont, Illinois
  - Springfield Clinic, Llp, Springfield, Illinois
  - Retina Associates of Kentucky, Lexington, Kentucky
  - Cumberland Valley Retina Consultants PC, Hagerstown, Maryland
  - Associated Retinal Consultants PC, Royal Oak, Michigan
  - Erie Retinal Surgery, Erie, Pennsylvania
  - Tennessee Retina PC, Nashville, Tennessee
  - Brown Retina Institute, San Antonio, Texas
  - Retina Center of Texas, Southlake, Texas
  - University of Utah, John Moran Eye Center, Salt Lake City, Utah
  - Piedmont Eye Center, Lynchburg, Virginia
  - Wagner Macula and Retina Center, Norfolk, Virginia
  - Spokane Eye Clinical Research, Spokane, Washington
- Argentina (5):
  - Salud Ocular, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto Oftalmologico de Buenos Aires S.A., Buenos Aires
  - Centro Oftalmologico Dr. Charles S.A., Ciudad Autonoma Buenos Aires
  - Centro Privado de Ojos Romagosa S.A, Córdoba
  - CEO Centro de Especialidades Oftalmologicas Tucuman, San Miguel de Tucumán
- Australia (8):
  - Retina and Macula Specialists, Hurstville, New South Wales
  - Sydney West Retina, Westmead, New South Wales
  - Sunshine Coast University Hospital, Geebung, Queensland
  - Centre For Eye Research Australia, East Melbourne, Victoria
  - Cabrini Hospital Malvern, Melbourne, Victoria
  - Retina Specialists Victoria, Rowville, Victoria
  - Lions Outback Vision Service in Broome, Broome, Western Australia
  - The Lions Eye Institute, Nedlands, Western Australia
- Bulgaria (5):
  - Medical Center for Eye Health ? Focus Ltd, Sofia
  - Specialized Eye Hospital Pentagram, Sofia
  - Specialized Hospital for Active Treatment of Ophthalmologic Diseases ?Zora?, OOD, Sofia
  - Eye Clinic St. Petka - Varna, Varna
  - SHEDAT - Varna EOOD, Varna
- Canada (11):
  - Retina Surgical Associates, New Westminster, British Columbia
  - Toronto Retina Institute, Don Mills, Ontario
  - St Joseph's Centre for Mountain Health Services, Hamilton, Ontario
  - St. Joseph's Health Care - London, London, Ontario
  - Retina Institute of Ottawa, Ottawa, Ontario
  - Clarity eye Institute, Vaughan, Ontario
  - Institut De L'Oeil Des Laurentides, Boisbriand, Quebec
  - Clinique d'ophtalmologie et de Retine de l'est, Montreal, Quebec
  - Eye Health MD (Opthalmology), Montreal, Quebec
  - Retina MD Clinic, Sainte-Catherine, Quebec
  - Centre Oculaire de Quebec, Québec
- Chile (2):
  - Red Salud UC Christus, Santiago, Santiago Metropolitan
  - Centro de la Vision, Las Condes
- Croatia (5):
  - General Hospital Karlovac, Karlovac
  - Clinical Hospital Centre Osijek, Osijek
  - Clinical Hospital Centre Rijeka, Rijeka
  - Special Hospital for Ophthalmology Svjetlost, Zagreb
  - University Hospital Center Zagreb, Zagreb
- Czechia (3):
  - Nemocnice Pardubickeho kraje a.s., Pardubice
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - Tomas Bata Regional Hospital, Zlín
- Denmark (3):
  - Ålborg Universitets Hospital, Aalborg
  - Rigshospitalet Glostrup, Glostrup Municipality
  - Sjllands Universitetshospital, Roskilde
- Egypt Air Hospital, Cairo, Egypt
- France (37):
  - Centre Ophtalmologique Maison-Rouge, Strasbourg, Bas Rhin
  - CH St Joseph, Marseille, Bouches Du Rh(ne
  - CHU Dijon - Hopital Francois Mitterrand, Dijon, Cte-d'Or
  - Groupe Hospitalier Pellegrin, Bordeaux, Gironde
  - CHU de Nantes - Hotel Dieu, Nantes, Loire Atlantique
  - Institut Ophtalmologique De l Ouest Jules Verne, Nantes, Paris
  - CHU de St-Etienne - Hopital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Hopital Edouard Herriot - CHU Lyon, Lyon, Rhone
  - Centre Hospitalier de la Croix Rousse, Lyon, Rhone
  - Clinique Mathilde, Rouen, Seine Maritime
  - Hopital Avicenne, Bobigny, Seine Saint Denis
  - CHU Amiens Picardie, Centre de Recherche Clinique, Amiens, Somme
  - Centre Hospitalier de Versailles, Le Chesnay, Yvelines
  - Aix Vision, Aix-en-Provence
  - Centre Rétine Gallien, Bordeaux
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Clinique du Val d'Ouest- Institut Rhône Alpin, Écully
  - Clinique des Yeux Bordeaux, Floirac
  - Centre d'Ophtalmologie, Fontainebleau
  - Centre Optha Du Dauphine, Grenoble
  - Hôpital Saint-Louis - La Rochelle, La Rochelle
  - Visiopole Private Practice, Lagord
  - Centre Ophtalmologique Rabelais, Lyon
  - Centre Ophtalmologique Kleber, Lyon
  - Centre Monticelli Paradis d Ophtalmologie, Marseille
  - Clinique de Montargis, Montargis
  - Clinique Honore Cave, Montauban
  - Alpes Retine, Montbonnot-Saint-Martin
  - Centre Des Arceaux, Montpellier
  - CHU Nice - Hôpital Saint Roch, Nice
  - Centre Ophtalmologique de L'Odeon, Paris
  - Centre Ophtalmologique d?Imagerie et de Laser, Paris
  - CHU Poitiers - Hôpital la Milétrie, Poitiers
  - Centre St Exupery, Saint-Cyr-sur-Loire
  - Institut Sourdille, Saint-Herblain
  - Clinique de l'Union, Saint-Jean
  - Chu Toulouse, Toulouse
- Germany (22):
  - Medical Eye Research Xpertx Institut gGmbH, Trier, Bavaria
  - Private Practice of Dr. Astrid Sader Moritz, Würzburg, Bavaria
  - Augenzentrum Prof. Koch GmbH, Frankfurt am Main, Hesse
  - Universitaetsklinikum Frankfurt Goethe-Universitaet, Frankfurt am Main, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitaetsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Apotheke am Klinikum Ludwigshafen, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Leipzig, Leipzig, Saxony
  - Augenzentrum Erzgebirge, Zschopau, Saxony
  - Martin-Luther-Universitaet Halle-Wittenberg - Staedtisches Klinikum Dessau (SKD), Dessau, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - St. Gertrauden Krankenhaus Berlin, Augenheilkunde, Berlin
  - Vivantes Klinikum Neukoelln, Berlin
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Halle (Saale), Halle
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Mannheim, Mannheim
  - Praxis Dr. Amin Gamael, Rostock
  - Universitaetsaugenklinik Rostock, Rostock
  - Knappschaftskrankenhaus Sulzbach, Sulzbach
- Hong Kong (2):
  - Grantham Hospital, Hong Kong
  - Hong Kong Eye Hospital, Kowloon
- Israel (7):
  - Rambam Health Care Campus, Haifa
  - Wolfson Medical Center, Holon
  - Hadassah, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin MC, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Hashalom Medical Center, Tel Aviv
- Italy (25):
  - Ospedale Clinicizzato SS. Annunziata, Chieti, Abruzzo
  - Azienda Ospedaliero Universitaria Consorziale Policlinico di Bari, Bari, Apulia
  - Azienda Ospedaliero Universitaria Mater Domini, Catanzaro, Calabria
  - Ospedale Monaldi - AORN dei Colli, Napoli, Campania
  - Azienda Ospedaliera di Udine Ospedale S. Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Fondazione Ptv Policlinico Tor Vergata, Rome, Lazio
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - G. B. Bietti Fondazione - IRCCS, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea-Universitr di Roma La Sapien, Rome, Lazio
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Humanitas Gavazzeni, Bergamo, Lombardy
  - Fondazione IRCCS CA? Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - Ospedale San Giuseppe Fatebenefratelli, Milan, Lombardy
  - Ospedale San Raffaele, Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Santi Paolo e Carlo (San Paolo-Polo Universitario), Milan, Lombardy
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli (Presidio Ospedale Sacco), Milan, Lombardy
  - Fondazione IRCCS - San Gerardo dei Tintori, Monza, Lombardy
  - Ente Ecclesiastico Ospedale Generale Regionale F Miulli, Acquaviva Delle Fonti, Piedmont
  - Ospedale Oftalmico, Turin, Piedmont
  - Città della Salute e della Scienza di Torino. Presidio Molinette, Turin, Piedmont
  - Ospedale Mauriziano Umberto I, Turin, Piedmont
  - Ospedale Di Sassuolo, Sassuolo, Sardinia
  - Azienda Ospedaliera Universitaria "Policlinico - Vittorio Emanuele" (Presidio Gaspare Rodolico), Catania, Sicily
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria delle Marche, Ancona, The Marches
- Japan (47):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - Nagoya University Hospital, Nagoya, Aichi-ken
  - Toho University Sakura Medical Center, Sakura-shi, Chiba
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe University Hospital, Kobe, Hyōgo
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Nihon University Hospital, Chiyoda-ku, Tokyo-To
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To
  - Chukyo Hospital, Aichi
  - Sugita Eye Hospital, Aichi
  - Nagoya City University Hospital, Aichi
  - Akita University Hospital, Akita
  - Chiba University Hospital, Chiba
  - Juntendo University Urayasu Hospital, Chiba
  - University of Yamanashi Hospital, Chuo-shi
  - Kyushu University Hospital, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Gifu University Hospital, Gifu
  - Hiroshima University Hospital, Hiroshima
  - Sapporo City General Hospital, Hokkaido
  - University of Tsukuba Hospital, Ibaraki
  - Kozawa eye hospital and diabetes center, Ibaraki
  - Kagawa University Hospital, Kagawa
  - NHO Tokyo Medical Center, Meguro-ku
  - Mie University Hospital, Mie
  - Fukushima Medical University Hospital, Miyagi
  - Shinshu University Hospital, Nagano
  - Nagasaki University Hospital, Nagasaki
  - Japanese Red Cross Nagasaki Genbaku Hospital, Nagasaki
  - Tazuke-kofukai Medical Research Institute Kitano Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Kansai Medical University Hospital, Osaka
  - Saitama Medical University Hospital, Saitama
  - Shiga University Of Medical Science Hospital, Shiga
  - Seirei Hamamatsu General Hospital, Shizuoka
  - Osaka University Hospital, Suita
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki-shi
  - Tokushima University Hospital, Tokushima
  - Juntendo University Hospital, Tokyo
  - Tokyo Women's Medical University Hospital, Tokyo
  - Kyorin University Hospital, Tokyo
  - Tokyo Medical University Hachioji Medical Center, Tokyo
  - Yamagata University Hospital, Yamagata
  - Yamaguchi University Hospital, Yamaguchi
  - University of Fukui Hospital, Yoshida-gun
- Poland (4):
  - Centrum Diagnostyki i Mikrochirurgii Oka LENS, Olsztyn
  - Szpital im. Jozefa Strusia, Poznan
  - Wojskowy Instytut Medyczny - Panstwowy Instytut Badawczy, Warsaw
  - Szpital Specjalistyczny im Soko?owskiego, Wałbrzych
- Emanuelli Research and Development Center, Arecibo, Puerto Rico
- King Khaled Eye Specialist Hospital, Riyadh, Saudi Arabia
- Singapore (5):
  - National University Hospital, Singapore
  - Singapore National Eye Centre, Singapore
  - Eye & Retina Surgeons, Singapore
  - Tan Tock Seng Hospital, Singapore
  - Eagle Eye Centre, Singapore
- Univerzitetni Klinicni Center Ljubljana Ocesna Klinika, Ljubljana, Slovenia
- South Korea (2):
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggi-do
  - Yeungnam University Hospital, Daegu
- Spain (25):
  - Hospital Universitari Son Espases, Palma de Mallorca, Balearic Islands
  - Fundacio Privada Hospital Asil de Granollers, Granollers, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Complejo Hospitalario Universitario de Ferrol, Ferrol, LA Coruna
  - Complejo Hospitalario Universitario de Santiago., Santiago de Compostela, LA Coruna
  - Complejo Hospitalario San Millán y San Pedro De La Rioja, Logroño, La Rioja
  - Hospital Universitario Insular de Gran Canaria, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Costa del Sol, Marbella, Malaga
  - Hospital Xeral-Cies de Vigo, Vigo, Pontevedra
  - Hospital Universitario Nuestra Señora de la Candelaria, Santa Cruz de Tenerife, Tenerife
  - Hospital de Basurto, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete, Albacete
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Dos de Maig, Barcelona
  - Hospital Universitari Vall dHebron (CEMCAT), Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Complejo Asistencial Universitario de Burgos, Burgos
  - Hospital Universitario Puerta del Mar, Cadiz
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen de Las Nieves, Granada
  - Hospital Carlos Haya, Málaga
  - Hospital Universitario Virgen de La Arrixaca, Murcia
  - Hospital Universitario Virgen Del Rocio Sevila, Seville
  - Hospital Universitario Rio Hortega, Valladolid
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (2):
  - Lund University Hospital, Lund
  - St Eriks Eye Hospital, Stockholm
- Switzerland (13):
  - Kantonsspital Aarau AG, Aarau
  - Universitätsspital Basel, Basel
  - Augenklinik am Lindenhofspital, Bern
  - Inselspital-Universitaetsspital Bern, Bern
  - Vista Augenklinik Binningen, Binningen
  - Hôpitaux Universitaires de Genève, Geneva
  - Hôpital ophtalmique Jules-Gonin, Lausanne
  - Swiss Visio Montchoisi, Lausanne
  - LUKS Spitalbetriebe AG, Lucerne
  - Ospedale Regionale di Lugano, Lugano
  - Pallas Klinik Olten, Olten
  - Kantonsspital St. Gallen, Sankt Gallen
  - Stadtspital Triemli, Zurich
- Taiwan (3):
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
  - Far Eastern Memorial Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District
- Thailand (7):
  - King Chulalongkorn Memorial Hospital, Pathum Wan, Bangkok
  - Srinagarind Hospital, Muang, Changwat Khon Kaen
  - Songklanagarind Hospital, Hat Yai, Changwat Songkhla
  - Metta Pracharak Hospital, Nakhon Pathom, RAI Khing
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital, Chiang Mai
- United Arab Emirates (3):
  - Burjeel Hopital, Abu Dhabi
  - Medcare Eye Center - Dubai, Dubai
  - Magrabi Eye Hospital, Dubai Healthcare City
- United Kingdom (28):
  - Bristol Eye Hospital, Bristol, Avon
  - Bedford Hospital, Bedford, Bedfordshire
  - Torbay Hospital, Torquay, Devon
  - Hull Royal Infirmary, Hull, East Riding Of Yorkshire
  - Primary Care Centre, Colchester, Essex
  - Gloucestershire Retinal Research Group, Gloucester, Gloucestershire
  - Kings College Hospital, London, Greater London
  - Maidstone Hospital, Maidstone, Kent
  - Royal Liverpool University Hospital, Liverpool, Merseyside
  - James Paget University Hospitals NHS Foundation Trust, Gorleston-on-Sea, Norfolk
  - John Radcliffe Hospital, Headington, Oxfordshire
  - Mater Infirmorum Hospital, Belfast
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Birmingham Midland Eye Centre, Birmingham
  - Bradford Royal Infirmary, Bradford
  - University Hospital of Wales, Cardiff
  - Frimley Park Hospital, Frimley
  - North West London Hospitals NHS Trust, Harrow
  - St James University Hospital, Leeds
  - Moorfields Eye Hospital, London
  - Royal Free Hospital, London
  - Manchester Royal Eye Hospital, Manchester
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - Sunderland Eye Infirmary, Sunderland
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing